CLINICAL TRIAL: NCT03491475
Title: Dynamicity of Echocardiography During Ajmaline Test
Brief Title: Echocardiography During Ajmaline Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Esther Scheirlynck, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: UniverstairZB
Record Dates: First submitted 2018-03-26; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Brugada Syndrome
Keywords: Ajmaline test
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negative Ajmaline test: No appearance of a type 1 ECG during Ajmaline test
  Interventions: Drug: Ajmaline test
- Positive Ajmaline test: Appearance of a type 1 ECG during Ajmaline test
  Interventions: Drug: Ajmaline test

INTERVENTIONS:
Drug: Ajmaline test — Administration of Ajmaline
  Other Names: Echocardiography

SUMMARY:
In this study the investigators analyse echocardiographic images before and during Ajmaline test. The purpose is to know if any echocardiographic modifications are present during either negative or positive Ajmaline testing.

DETAILED DESCRIPTION:
The diagnosis of Brugada Syndrome is made when a type 1 pattern is present on the electrocardiogram (ECG), either spontaneously or after administration of a sodium channel blocker. For pathofysiological understanding, the investigators will analyse echocardiography images before and during the administration of Ajmaline. Comparing echocardiographies before and during negative Ajmaline test, will allow the investigators to indentify the effect of Ajmaline administration on cardiac function. The comparison between images of negative and positive Ajmaline tests will expose differences related to the occurence of a type 1 ECG.

ELIGIBILITY:
Inclusion Criteria:

* >17 years old
* clinical indication for Ajmaline test

Exclusion Criteria:

* History of right ventricular outflow tract ablation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for Ajmaline test, either because of symptoms or in the context of familial screening.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Speckle tracking strain measurement | 1 day at the time of enrollment
  Cardiac function assessed by speckle tracking peak strain and peak strain dispersion

CONTACTS AND LOCATIONS:
Overall Officials: Esther Scheirlynck, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided